CLINICAL TRIAL: NCT03855423
Title: Malaysian Tocotrienol Rich Fraction: Immunomodulatory Effect in Women With Breast Cancer
Brief Title: Maximum Tolerated Dose, Safety and Pharmacologic Study of TRF in Women With Breast Cancer
Acronym: Matriac
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nur Aishah Mohd Taib (Other)
Collaborators: Malaysia Palm Oil Board (Other Government)
Responsible Party: Sponsor-Investigator, Nur Aishah Mohd Taib, Professor, University of Malaya
Organization: University of Malaya (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 853.4
Record Dates: First submitted 2019-02-14; First posted 2019-02-26 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer Female
Keywords: MTD; TRF; Pharmacology

STUDY DESIGN:
Intervention Model Description: Single arm intervention study 3+3 step up design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocotrienol-rich Fraction (TRF) (Experimental): Pre-operative patients will be receiving TRF at different doses assigned to them in a cohort of 3 patients at each level.
  Interventions: Dietary Supplement: Tocotrienol-rich Fraction (TRF)

INTERVENTIONS:
Dietary Supplement: Tocotrienol-rich Fraction (TRF) — TRF consists of alpha, gamma and delta tocotrienols in addition to small amount of alpha-tocopherol
  Other Names: Tocovid Suprabio

SUMMARY:
Phase Ib: Maximum Tolerated Dose, Safety and Pharmacologic Study of TRF in Women with Breast Cancer is aimed to determine the highest, safest and tolerable dose of Tocotrienol-rich Fraction (maximal tolerated dose: MTD) that can be used in women with breast cancer.

DETAILED DESCRIPTION:
3+3 step up design method will be used in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with operable breast cancer
* Life expectancy of at least 3 months
* Adequate organ function
* No allergy to Vitamin E and TRF
* Provides consent to participate in trial and adhere to the study protocol

Exclusion Criteria:

* Receiving concomitant chemotherapy, radiotherapy, hormonal, immune therapy or other investigational drugs
* Uncontrolled concurrent illness
* Pregnant / breast feeding women
* Patients who are unable or unwilling to take Tocotrienols, herbal remedies, or non-prescription medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Assessment | For 2 to 4 weeks during supplementation
  Number of participants with treatment-related adverse events as assessed by CTCAE version 5.0
Liver Function Test | For 2 to 4 weeks during supplementation
  Liver enzymes with units of U/L

SECONDARY OUTCOMES:
Bioavailability of TRF | For 2 to 4 weeks during supplementation
  Blood pharmacokinetic parameters

CONTACTS AND LOCATIONS:
Overall Officials: Nur Aishah Taib, MBBS, Principal Investigator — University of Malaya
Locations (1):
- University of Malaya Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No